CLINICAL TRIAL: NCT01308333
Title: Investigation of Chronic Inflammatory Processes in the Respiratory Tract and the Eyes of Male Individuals With X-linked Hypohidrotic Ectodermal Dysplasia
Brief Title: Investigation of Chronic Inflammatory Processes in Male Individuals With Hypohidrotic Ectodermal Dysplasia
Status: Completed | Type: Observational
Sponsor: University Hospital Erlangen (Other)
Collaborators: Edimer Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Prof. Dr. Holm Schneider, Head of the Division of Molecular Pediatrics, University Hospital Erlangen
Other Study IDs: ED11
Record Dates: First submitted 2011-03-03; First posted 2011-03-04 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2014-01

CONDITIONS: X-linked Hypohidrotic Ectodermal Dysplasia
MeSH Terms: conditions — Ectodermal Dysplasia 1, Anhidrotic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — tear fluid

GROUPS / COHORTS (4):
- XLHED children
- XLHED adults
- Control children
- Control adults

SUMMARY:
X-linked hypohidrotic ectodermal dysplasia (XLHED) is a complex genetic disorder characterized by lack of sweat, sebaceous, submucous, Meibomian and mammary glands, sparse hair and eyebrows, and oligodontia. Insufficient function of the respective glands may lead to chronic inflammatory processes in airways and eyes of the affected individuals. The investigators will quantify sweat glands of XLHED patients, assess chronic conjunctivitis and blepharitis in conjunction with quantitative and/or qualitative alterations of lacrimal fluid in these subjects, evaluate lung function and assess chronic inflammatory processes in the airways by NO measurements. The data should provide a basis for genotype-phenotype correlations.

ELIGIBILITY:
Inclusion Criteria:

* for patients: X-linked hypohidrotic ectodermal dysplasia caused by mutations in the gene EDA
* written informed consent

Exclusion Criteria:

* acute respiratory disease
* acute allergic problem, e.g. allergic coryza
* implantable electronic devices, e.g. pacemaker

Ages: 6 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: subjects with X-linked hypohidrotic ectodermal dysplasia (XLHED) and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2011-04; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holm Schneider, MD, Principal Investigator — University Hospital Erlangen
Locations (1):
- University Hospital Erlangen, Competence Centre for Children with Ectodermal Dysplasias, Erlangen, Bavaria, Germany

REFERENCES:
- [Result] Dietz J, Kaercher T, Schneider AT, Zimmermann T, Huttner K, Johnson R, Schneider H. Early respiratory and ocular involvement in X-linked hypohidrotic ectodermal dysplasia. Eur J Pediatr. 2013 Aug;172(8):1023-31. doi: 10.1007/s00431-013-1985-8. Epub 2013 Apr 4. PMID 23553579